CLINICAL TRIAL: NCT03327051
Title: The Effect of Gastric Acid Suppression on Probiotic Colonization
Brief Title: Gastric Acid Suppression and Probiotic Colonization
Acronym: PR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Aida Habtezion, Associate Professor of Medicine (Gastroenterology and Hepatology), Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 41681
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Results first posted 2020-01-07 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Probiotics
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Omeprazole and VSL #3 (Active Comparator): Participants will receive a proton pump inhibitor (Omeprazole) and VSL #3 Probiotics
  Interventions: Drug: Omeprazole; Dietary Supplement: VSL #3
- Placebo and VSL #3 (Placebo Comparator): Participants will receive placebo and VSL #3 Probiotics
  Interventions: Dietary Supplement: VSL #3; Drug: Placebo

INTERVENTIONS:
Drug: Omeprazole — Proton pump inhibitor (PPI) that suppresses gastric acid secretion
  Arms: Omeprazole and VSL #3
Dietary Supplement: VSL #3 — Probiotics
Drug: Placebo — Placebo to match omeprazole
  Arms: Placebo and VSL #3

SUMMARY:
Probiotics are over-the-counter dietary products with microorganisms that are generally consumed for health benefit. However, the durability of these microorganisms is unclear, particularly when they pass through the highly acidic environment of the stomach. We will test the colonization of these microorganisms among individuals who consume probiotics with and without acid suppression therapy.

DETAILED DESCRIPTION:
All activities will be related to research. Participants will be randomized to receive either over-the-counter acid suppression medication or placebo from weeks -2 through week 4. All participants will receive VSL #3 (over-the-counter probiotic) from weeks 0 through 4. Survey data, serum, and stool samples will be collected at weeks -2, 0, and 4.

The intervention medication and probiotics have a very low side effect profile and are available over the counter. All data collection methods are non-invasive.

Elucidation of the effects of acid suppression on probiotic colonization will allow us to better understand the utility of probiotics use by individuals on acid suppression medications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ages 18 years and ≤ 75 years.
* Able to visit the study Doctor's office 3 times, answer 3 questionnaires, and provide stools and blood samples.

Exclusion Criteria:

* Gastric cancer, Barrett's esophagus cancer, any gastrointestinal condition, or soy or gluten sensitivity
* Previous abdominal surgery
* Currently pregnant or nursing
* Had H. Pylori Infection
* Diagnosed with any chronic medical condition other than hypertension or hyperlipidemia
* Currently consuming herbs or probiotics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aida Habtezion, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh G, Haileselassie Y, Briscoe L, Bai L, Patel A, Sanjines E, Hendler S, Singh PK, Garud NR, Limketkai BN, Habtezion A. The effect of gastric acid suppression on probiotic colonization in a double blinded randomized clinical trial. Clin Nutr ESPEN. 2022 Feb;47:70-77. doi: 10.1016/j.clnesp.2021.11.005. Epub 2021 Nov 10. PMID 35063245

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants attended an initial study visit at week -2, followed by a baseline visit at week 0, and a final visit at week 4.
Groups:
- Omeprazole and VSL #3: Proton pump inhibitor (Omeprazole) and VSL #3 Probiotics
- Placebo and VSL #3: Placebo and VSL #3 Probiotics
Period: Overall Study
Arm/Group | Omeprazole and VSL #3 | Placebo and VSL #3
Started | 19 | 20
Received Treatment | 16 | 16
Attended Visit 2 (Week 0) | 15 | 15
Completed | 14 | 15
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were collected at visit 2 (week 0). Participants who attended visit 2 are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omeprazole and VSL #3 | Placebo and VSL #3 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (13) | 37 (12) | 37 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 4 | 6 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic / White | 3 | 2 | 5
  Hispanic / Other | 2 | 1 | 3
  NonHispanic / White | 7 | 6 | 13
  NonHispanic / Other | 0 | 1 | 1
  NonHispanic / Asian | 2 | 4 | 6
  NonHispanic / Black or African American | 1 | 0 | 1
  NonHispanic / Native Hawaiian / Pacific Islander | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Relative Abundance of Probiotic Strains [Mean (Standard Deviation); unit: percentage of abundance] — Relative abundance is reported as the percent of combined probiotic strains in the bacteria sample (S. thermophiles, B. breve, B. longum, B. infantis, L. acidophilus, L. plantarum, L. paracasei, L. delbrueckii subsp. bulgaricus).
  percentage of abundance | 0.3653 (0.407) | 0.5875 (0.5691) | 0.4764 (0.4907)
Number of participants experiencing gastro-intestinal symptoms. [Count of Participants; unit: Participants] — Participants were asked to report symptoms of gastro-intestinal discomfort experienced within the last 28 days.
  Participants
    Bloating | 1 | 3 | 4
    Flatulence | 1 | 0 | 1
    Diarrhea | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Relative Abundance of VSL#3 Probiotic Bacterial Strains When Ingested in the Presence or Absence of the Proton Pump Inhibitor (PPI) Omeprazole at Week 4.
Description: Relative abundance is reported as the percent of combined VSL #3 probiotic bacteria strains in the bacteria sample (S. thermophiles, B. breve, B. longum, B. infantis, L. acidophilus, L. plantarum, L. paracasei, L. delbrueckii subsp. bulgaricus) following their ingestion in the presence or absence of the gastric acid suppression drug omeprazole. Stool samples were assessed.
Time Frame: Week 4
Population: Participants who attended the week 4 visit are included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of abundance
Arm/Group | Omeprazole and VSL #3 | Placebo and VSL #3
Number analyzed (Participants) | 14 | 15
percentage of abundance | 1.002 (0.8403) | 0.8186 (0.5234)
Statistical Analysis 1: Comparison: Omeprazole and VSL #3; Within group difference between week 0 and week 4 was analyzed; Test type: Other — An increase in relative abundance of VSL3 bacterial strains at week 4 compared to week 0 (baseline) is considered significant if p<0.05; p = 0.04, ANOVA; Two-way ANOVA with Bonferroni post-test was used for multi-variable analysis
Statistical Analysis 2: Comparison: Placebo and VSL #3; Within group difference between week 0 and week 4 was analyzed; Test type: Other — [test comment as in outcome 1, analysis 1]; p > 0.99, ANOVA; Two-way ANOVA with Bonferroni post-test was used for multi-variable analysis

2. Secondary Outcome: Number of Participants With Symptoms Related to VSL#3 Treatment.
Description: Participants were asked to report symptoms of gastro-intestinal discomfort experienced within the last 28 days.
Time Frame: Week 0 through Week 4
Population: Participants who attended the week 4 visit are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Omeprazole and VSL #3 | Placebo and VSL #3
Number analyzed (Participants) | 14 | 15
Participants
  Bloating | 0 | 2
  Flatulence | 2 | 0
  Diarrhea | 2 | 0

3. Secondary Outcome: Relative Abundance (Mean Value) of Most Abundant Bacterial Phylum Before and After VSL#3 Probiotic Administration
Description: From week 0 to week 4, change in the relative abundance (percentage) of most common types of bacteria phyla normally found in the lower GI track (e.g. Firmicutes, Bacteroidetes, Actinobacteria and Proteobacteria) after ingesting VSL#3 in the presence or absence of omeprazole. Stool samples are assessed.
Time Frame: Week 0 and Week 4
Population: Participants who attended the week 4 visit are included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of abundance
Arm/Group | Omeprazole and VSL #3 | Placebo and VSL #3
Number analyzed (Participants) | 14 | 15
percentage of abundance
  Bacteroidetes at Week 0 | 66.4 (15.1) | 65.6 (11.3)
  Bacteroidetes at Week 4 | 66.2 (15.0) | 68.1 (10.2)
  Firmicutes at Week 0 | 25.6 (9.6) | 27.2 (9.6)
  Firmicutes at Week 4 | 25.7 (12.6) | 25.0 (8.3)
  Proteobacteria at Week 0 | 4.1 (6.0) | 2.7 (1.8)
  Proteobacteria at Week 4 | 3.12 (3.7) | 2.7 (2.4)
  Actinobacteria at Week 0 | 2.5 (2.5) | 3.2 (2.8)
  Actinobacteria at Week 4 | 3.7 (3.7) | 3.2 (1.9)

4. Secondary Outcome: Change in Peak Intensity of the Metabolite 1H-Indole-4-carbaldehyde Before and After VSL#3 Probiotic Administration (Omeprazole and VSL #3).
Description: From week 0 to week 4, relative change in metabolites (e.g. short chain fatty acids, bile acid derivatives, flavonoids, amino acids) found in the GI track by mass spectrometry after ingesting VSL#3. Serum samples are assessed.
  MZ = mass/charge ratio; RT = retention time. MZ/RT data were obtained by mass spectrometry analysis. This is a metabolite of interest for the Omeprazole and VSL#3 group only.
Time Frame: Week 0 and Week 4
Population: Participants in the Omeprazole and VSL#3 group who attended the week 4 visit are included in the analysis.
Measure: Mean (Standard Deviation); unit: MZ/RT
Arm/Group | Omeprazole and VSL #3
Number analyzed (Participants) | 14
MZ/RT
  1H-Indole-4-carbaldehyde at Week 0 | 80809.5 (118044.6)
  1H-Indole-4-carbaldehyde at Week 4 | 286707.9 (567693.1)

5. Secondary Outcome: Change in Peak Intensity of Metabolites of Interest Before and After VSL#3 Probiotic Administration (Placebo and VSL#3 Group).
Description: From week 0 to week 4, relative change in metabolites (e.g. short chain fatty acids, bile acid derivatives, flavonoids, amino acids) found in the GI track by mass spectrometry after ingesting VSL#3. Serum samples are assessed.
  MZ = mass/charge ratio; RT = retention time. MZ/RT data were obtained by mass spectrometry analysis. These are metabolites of interest for the Placebo and VSL#3 group only.
Time Frame: Week 0 and Week 4
Population: Participants in the Placebo and VSL#3 group who attended the week 4 visit are included in the analysis.
Measure: Mean (Standard Deviation); unit: MZ/RT
Arm/Group | Placebo and VSL #3
Number analyzed (Participants) | 15
MZ/RT
  11-OXOURSOLIC ACID ACETATE at Week 0 | 95819.8 (146506.5)
  11-OXOURSOLIC ACID ACETATE at Week 4 | 4726.2 (18243.3)
  FA(14:0) at Week 0 | 539032.9 (519162.2)
  FA(14:0) at Week 4 | 249632.3 (219622.8)
  Iloprost S-isomer at Week 0 | 87765.6 (189360.0)
  Iloprost S-isomer at Week 4 | 22405.5 (63899.1)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Omeprazole and VSL #3 | Placebo and VSL #3
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 7/19 | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omeprazole and VSL #3 (N=19) | Placebo and VSL #3 (N=20)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 2 (2)
Increased stool frequency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 4 (7)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT03327051/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT03327051/SAP_001.pdf